CLINICAL TRIAL: NCT06412835
Title: The Effect of Cooperative Learning Approach on Nursing Students' Learning of Knowledge and Skills Regarding Enteral Nutrition: a Randomized Controlled Study
Brief Title: Enteral Nutrition Training with Cooperative Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bilecik Seyh Edebali Universitesi (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: Aysun Acun 6
Record Dates: First submitted 2024-05-03; First posted 2024-05-14 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-05

CONDITIONS: Educational Problems
Keywords: cooperative learning; nursing students; enteral nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Students' course success (Experimental): Knowledge level of nursing students
  Interventions: Other: cooperative learning
- self-directed learning (Experimental): self-directed learning
  Interventions: Other: cooperative learning

INTERVENTIONS:
Other: cooperative learning — Students working in groups

SUMMARY:
Nursing students; education on enteral nutrition has an important place. With cooperative learning, students will make their learning permanent by communicating with each other. This study is carried out to evaluate the effect of cooperative learning on the knowledge level of students.

DETAILED DESCRIPTION:
The cooperative learning method is structured on students' communication and interaction with each other. Many outcomes such as increasing students; academic success, critical thinking, verbal communication, taking responsibility for learning, improving their ability to take responsibility, increasing their ability to evaluate, and being open to feedback are among the benefits of cooperative learning. In cooperative learning, the basic principle is that students form groups and share their knowledge within each group regarding the basic knowledge and skills they want to learn, and then the groups interact with each other. With this method, students can take on learning responsibilities themselves, and they can also develop their knowledge sharing, collaboration and leadership skills within the group. Therefore, cooperative learning is an effective training method by strengthening self-directed learning, as well as supporting effective communication within team members. In a study conducted with nursing students using cooperative learning, it was observed that higher success, more positive relationships between students, and more psychological adaptation developed compared to traditional education methods. In international studies investigating the use of active learning strategies in nursing education, it has been concluded that collaborative learning is of great importance in transforming critical thinking ability, clinical performance, knowledge adequacy and nursing knowledge into clinical skills. In a similar vein, it has been emphasized that cooperative learning is an effective teaching method in improving the knowledge and psychomotor skill levels of nursing students regarding local drug applications and increasing the permanence of information. This study will focus on students; learning of knowledge and skills regarding enteral nutrition through cooperative learning method. A more memorable learning is aimed by students forming groups and transferring information both within and between groups.

ELIGIBILITY:
Inclusion Criteria:

* Getting training on enteral nutrition for the first time
* Volunteering to participate in the study
* Being required to attend class

Exclusion Criteria:

* Having previously received training on enteral nutrition
* Not volunteering to participate in the study
* Not participating in the final test and follow-up test

Ages: 17 Years to 37 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2024-05-08 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-06-07 (Actual)

PRIMARY OUTCOMES:
Knowledge level of nursing students | 5 weeks for each participant
  Nursing students' knowledge levels will be evaluated at the end of the teaching with the cooperative learning model on enteral nutrition.

CONTACTS AND LOCATIONS:
Locations (1):
- Bilecik Şeyh Edebali University, Bilecik, Bilecik, Turkey (Türkiye)